CLINICAL TRIAL: NCT01906268
Title: Attentional Bias Modification Treatment (ABMT) as Adjuvant Therapy for Anxiety Disorder Patients Resistent to Antidepressants: A Randomized Clinical Trial
Brief Title: Attention Retraining for Anxiety Disorder Patients Resistent to Antidepressants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-0338
Record Dates: First submitted 2013-07-08; First posted 2013-07-24 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder
Keywords: Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Antidepressants Resistant; Attentional Bias Modification Treatment (ABMT); Attentional Retraining; Adjuvant Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Panic Disorder | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- TAU + ABMT active (Experimental): Treatment as usual (TAU): selective serotonin reuptake inhibitor or serotonin-noradrenaline reuptake inhibitor
  Attention Bias Modification Treatment (ABMT) - active
  Interventions: Other: Attentional Bias Modification Treatment (ABMT) - Active
- TAU + AMBT placebo (Sham Comparator): Treatment as usual (TAU): selective serotonin reuptake inhibitor or serotonin norepinephrine reuptake inhibitor
  Attention Bias Modification Treatment (ABMT) - placebo (sham)
  Interventions: Other: Attentional Bias Modification Treatment - Placebo

INTERVENTIONS:
Other: Attentional Bias Modification Treatment (ABMT) - Active — The ABMT consists of 160 trials (120 angry-neutral and 40 neutral-neutral presentations). In the ABM condition, the target appears at the neutral-face location in all angry-neutral trials. Probe type (< or >) is not factorially counterbalanced but appears with equal probability for each of the following: angry-face location, probe location, or actor.
  Number of sessions: 10 ABMT sessions, 5 weeks (2 sessions once a week occurring in the same day with 40 minutes interval)
  Arms: TAU + ABMT active
Other: Attentional Bias Modification Treatment - Placebo — The Placebo protocol consists of 160 trials (120 angry-neutral and 40 neutral-neutral presentations). In the placebo condition, angry-face location, probe location, and actor are fully counterbalanced in presentation.
  Number of sessions: 10 ABMT sessions, 5 weeks (2 sessions once a week occurring in the same day with 40 minutes interval)
  Arms: TAU + AMBT placebo

SUMMARY:
The objective of this project is to test the combination of active or placebo Attentional Bias Modification Treatment (ABMT) to usual treatment for anxiety disorder patients resistant to antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Generalized Anxiety Disorder, Panic Disorder or Social Anxiety Disorder according to the International Neuropsychiatric Interview psychiatric interview (M.I.N.I.)
* Current treatment for the anxiety disorder with antidepressants with an appropriate dose for at least 8 weeks;
* Score on OASIS (Overall Anxiety Severity and Impairment Scale)equal or greater than 8

Exclusion Criteria:

* Other psychiatric disorder that causes more impairment and suffering than generalized anxiety disorder, panic disorder or social anxiety disorder in the clinical evaluation
* Current Cognitive Behavior Therapy
* Marked intellectual disability (clinically evident)
* Suicidal ideation or suicide plan at the time of assessment(M.I.N.I.)
* Psychotic disorder (M.I.N.I.)
* Bipolar disorder type I (M.I.N.I.)
* Abuse / Dependence substances (M.I.N.I.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale (OASIS) | Endpoint and 3-months follow-up
  Disorder non-specific primary outcome:
  Score change on OASIS (Overall Anxiety Severity and Impairment Scale) from baseline to endpoint and 3-months follow-up
Panic Disorder Severity Scale (PDSS), Generalized Anxiety Disorder 7-item Scale (GAD-7) or Liebowitz Social Anxiety Scale (LSAS) | Endpoint and 3-months follow up
  Disorder-specific primary outcome:
  For patients with Panic Disorder - change from baseline to endpoint and 3 months follow-up in the PDSS
  For patients with Generalized Anxiety Disorder - change from baseline to endpoint and 3 months follow-up in the GAD-7
  For patients with Social Anxiety Disorder - change from baseline to endpoint and 3 months follow-up in the LSAS

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Endpoint and 3-months follow-up
  Score change on BDI from baseline to endpoint and 3-months follow up
Beck Anxiety Inventory (BAI) | Endpoint and 3-months follow-up
  Score change on BAI from baseline to endpoint and 3-months follow up
DSM-5 Cross-Disorder Dimensional Scale [Brazilian version] | Endpoint and 3-months follow-up
  Score change on Cross-D from baseline to endpoint and 3-months follow up
Profile of Mood States (POMS) | Endpoint and 3-months follow-up
  Score Change on POMS from baseline to endpoint and 3-months follow up.
Clinical Global Impression(CGI) | Endpoint and 3-months follow-up
  Dichotomous outcome: percentage of patients with a score of 2 or less at the endpoint and 3-months follow-up evaluations

OTHER OUTCOMES:
Dot-probe and Executive Function Measures | Endpoint and 3-months follow-up
  Change in bias in attention orienting and executive function measures from baseline to endpoint and 3-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gisele G Manfro, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil